CLINICAL TRIAL: NCT06676293
Title: Compassionate Use of Combination Therapy with Asparaginase and Pembrolizumab in Patients with Nasopharyngeal Carcinoma
Brief Title: Compassionate Use of Asparaginase and Pembrolizumab Combination Theaapy for Nasopharyngeal Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB NO. 202400085B0
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Nasopharyngeal Carcinoma (NPC)
Keywords: NPC; ICB; asparaginase
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — spartalizumab; Asparaginase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- combination therapy (Experimental): The patients will receive asparaginase 10000IU/vail IM QD for three or five days, followed by pembrolizumab treatment. and Pembrolizumab 100mg in normal saline 100ml infusion over 30 minutes.
  Interventions: Drug: Anti-PD1; Drug: asparaginase
- anti-PD1 alone (Placebo Comparator): The patients will receive pembrolizumab treatment.
  Interventions: Drug: Anti-PD1

INTERVENTIONS:
Drug: Anti-PD1 — Pembrolizumab 100mg in normal saline 100ml infusion over 30 minutes for every two month
Drug: asparaginase — The patients will receive asparaginase 10000IU/vail IM QD for three or five days.
  Arms: combination therapy

SUMMARY:
The goal of this study is to investigate the outcomes of patients with locoregionally advanced nasopharyngeal carcinoma (LA-NPC) or recurrent-metastatic nasopharyngeal carcinoma (RM-NPC) treated with a combination of immune checkpoint blockade (ICB) and asparaginase.

DETAILED DESCRIPTION:
This study is being conducted to investigate the synergistic effect of combining asparaginase with immune checkpoint blockade (ICB) in tumor-bearing mice. Findings indicate that asparaginase enhances CD8+ T cell activation, and previous reports have shown that nasopharyngeal carcinoma (NPC) patients exhibit a lower response rate to ICB treatment. This study aims to determine whether the combination therapy of asparaginase and ICB is more effective or less effective compared to the standard ICB-only approach for patients with locoregionally advanced (LA-NPC) or recurrent-metastatic NPC (RM-NPC). Participants are being enrolled who have previously received ICB but continue to experience disease progression.

ELIGIBILITY:
Inclusion Criteria: Patients who have previously received immune checkpoint blockade therapy but are still experiencing disease progression -

Exclusion Criteria: Active autoimmune disease

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Quantitative Analysis of Plasma EBV DNA Levels for Treatment Response | Until the end of the study
  In nasopharyngeal carcinoma (NPC), plasma Epstein-Barr virus (EBV) DNA serves as a crucial biomarker for both diagnosis and monitoring. EBV, a herpesvirus that infects epithelial cells, is strongly associated with NPC development, especially in endemic regions. The transformation from latent EBV infection to active viral replication is considered a critical step in NPC pathogenesis. This transformation can be detected through circulating viral DNA levels in plasma or by measuring antibodies against various EBV antigens, such as EBNA1, VCA, and EA-D. Elevated EBV DNA levels often correlate with tumor burden and may serve as a predictor of NPC recurrence or progression. Consequently, plasma EBV DNA testing has become an essential tool in NPC clinical management, helping to guide treatment decisions and evaluate treatment response.

SECONDARY OUTCOMES:
FDG PET/CT scan | 3 month
  FDG PET/CT for detecting tumor existence

CONTACTS AND LOCATIONS:
Overall Officials: Huang-Yu Yang, M.D./Ph.D, Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan, Taiwan

REFERENCES:
- [Background] Gnanaprakasam JNR, Kushwaha B, Liu L, Chen X, Kang S, Wang T, Cassel TA, Adams CM, Higashi RM, Scott DA, Xin G, Li Z, Yang J, Lane AN, Fan TW, Zhang J, Wang R. Asparagine restriction enhances CD8+ T cell metabolic fitness and antitumoral functionality through an NRF2-dependent stress response. Nat Metab. 2023 Aug;5(8):1423-1439. doi: 10.1038/s42255-023-00856-1. Epub 2023 Aug 7. PMID 37550596